CLINICAL TRIAL: NCT06642493
Title: Efficacy of Fresh Frozen Plasma (Ffp) in the Treatment of Thrombocytopenia in Dengue Patients
Brief Title: Efficacy of Fresh Frozen Plasma (FFP) in Treating Thrombocytopenia in Dengue Patients
Acronym: EFFP-TDP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheikh Hasina National Institute of Burn and Plastic Surgery (Other)
Responsible Party: Principal Investigator, Ashraful Hoque, Assistant Professor, Sheikh Hasina National Institute of Burn and Plastic Surgery
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: SHNIBPS: June2024/03
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
Keywords: Dengue fever; Thrombocytopenia; Plasma transfusion; Elevated aPTT; Coagulopathy in dengue; Non-bleeding dengue complications; Hemostatic management in dengue
MeSH Terms: conditions — Dengue; Severe Dengue; Thrombocytopenia

STUDY DESIGN:
Intervention Model Description: In this model, participants are randomly assigned to one of two or more groups (arms) simultaneously, with each group receiving a different intervention or control treatment. The outcomes of each group are then compared to assess the efficacy and safety of the interventions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Intervention Arm Title: Plasma Transfusion. (Experimental): Arm 1: Intervention Arm Title: Plasma Transfusion Description: Participants in this arm will receive fresh frozen plasma (FFP) transfusion at a dose of 10-15 mL/kg body weight.
  Intervention:
  Type: Biological Name: Fresh Frozen Plasma (FFP) Description: Administration of FFP to correct coagulopathy and normalize aPTT.
  Interventions: Biological: Fresh frozen plasma
- Arm 2: Control Arm Title: Standard Supportive Care (Placebo Comparator): Arm 2: Control Arm Title: Standard Supportive Care Description: Participants in this arm will receive standard supportive care without plasma transfusion.
  Intervention:
  Type: Other Name: Standard Supportive Care Description: Standard medical management without the administration of plasma transfusion.
  Interventions: Biological: Fresh frozen plasma

INTERVENTIONS:
Biological: Fresh frozen plasma — Intervention Type: Biological
  * Intervention Name: Fresh Frozen Plasma (FFP)
  * Detailed Description:
  * Dosage:Fresh frozen plasma (FFP) will be administered at a dose of 10-15 mL/kg body weight.
  * Administration: The FFP will be transfused intravenously under controlled clinical conditions.
  * Purpose: The transfusion aims to correct coagulopathy and normalize activated partial thromboplastin time (aPTT) in non-bleeding thrombocytopenic dengue patients.
  * Monitoring: Patients will be closely monitored for any adverse reactions or complications during and after the transfusion process. Coagulation parameters, including aPTT, will be measured at baseline, 24 hours, and 48 hours post-transfusion.

SUMMARY:
This clinical trial seeks to assess the effectiveness of fresh frozen plasma (FFP) in the treatment of thrombocytopenia in individuals with dengue. Dengue is a viral infection marked by thrombocytopenia, potentially resulting in significant hemorrhagic consequences. FFP is frequently utilized in the management of coagulopathies, and this study will investigate its efficacy in enhancing platelet count and mitigating bleeding risks in dengue patients with thrombocytopenia. The research will be executed as a randomized, controlled trial to evaluate outcomes in patients receiving routine care with and without FFP transfusion.

DETAILED DESCRIPTION:
Background:

Dengue fever is a mosquito-borne viral disease prevalent in tropical and subtropical regions. Severe dengue can lead to complications such as thrombocytopenia (low platelet count) and coagulopathy, indicated by prolonged activated partial thromboplastin time (aPTT). While platelet transfusions are commonly used to manage thrombocytopenia, the potential benefits of plasma transfusion in non-bleeding thrombocytopenic dengue patients with elevated aPTT remain unexplored. Plasma contains essential coagulation factors that might normalize aPTT and stabilize the hemostatic system, preventing progression to bleeding episodes.

Hypothesis:

Plasma transfusion in non-bleeding thrombocytopenic dengue patients with elevated aPTT will improve coagulation parameters and reduce the risk of bleeding complications.

Objectives:

1. Assess the effect of plasma transfusion on aPTT in non-bleeding thrombocytopenic dengue patients.
2. Evaluate the clinical outcomes, including the incidence of bleeding complications, in patients receiving plasma transfusion.
3. Determine the safety and feasibility of plasma transfusion in this patient population.
4. Measure changes in other coagulation parameters such as prothrombin time (PT) and fibrinogen levels post-transfusion.
5. Observe overall clinical outcomes, including the length of hospital stay and mortality rates.

Study Design:

This is a randomized controlled trial (RCT) involving non-bleeding thrombocytopenic dengue patients with elevated aPTT.

Study Population:

* Inclusion Criteria:** Patients diagnosed with dengue fever, thrombocytopenia (platelet count < 50,000/μL), and elevated aPTT (> 40 seconds) without active bleeding.
* Exclusion Criteria: Patients with active bleeding, known coagulopathies unrelated to dengue, or contraindications to plasma transfusion.

Sample Size:

A total of 300 patients will be recruited. 150 patients will be assigned to the intervention group (receiving plasma transfusion) and 150 patients to the control group (receiving standard supportive care).

Intervention:

Patients in the intervention group will receive fresh frozen plasma (FFP) transfusion at a dose of 10-15 mL/kg body weight. The control group will receive standard supportive care without plasma transfusion.

Outcome Measures:

* Primary Outcome: Change in aPTT values from baseline to 24 and 48 hours post-transfusion.
* Secondary Outcomes: Incidence of bleeding complications within 7 days post-transfusion, changes in other coagulation parameters (PT, fibrinogen levels) from baseline to 24 and 48 hours post-transfusion, platelet count changes post-transfusion, length of hospital stay, and overall mortality rate within 30 days.

Data Collection:

Blood samples will be collected at baseline, 24 hours, and 48 hours post-transfusion to measure aPTT and other coagulation parameters. Clinical data, including bleeding episodes and other adverse events, will be recorded throughout the hospital stay.

Statistical Analysis:

Data will be analyzed using appropriate statistical methods. Continuous variables will be compared using t-tests or Mann-Whitney U tests, while categorical variables will be compared using chi-square tests. A p-value of < 0.05 will be considered statistically significant.

Ethical Considerations:

The study will be conducted in accordance with the Declaration of Helsinki and will be approved by the institutional ethics committee. Informed consent will be obtained from all participants or their legal guardians.

Expected Outcomes:

It is anticipated that plasma transfusion will normalize aPTT and improve coagulation parameters in non-bleeding thrombocytopenic dengue patients, thereby reducing the risk of bleeding complications and improving overall clinical outcomes.

Timeline:

* Study Design and Ethical Approval: 1 month
* Patient Recruitment and Data Collection: 3 months
* Data Analysis and Interpretation: 1 month
* Manuscript Preparation and Submission: 1 month

Budget:

The budget will cover the costs of plasma units, laboratory tests, personnel salaries, and other administrative expenses. A detailed budget will be provided upon approval of the proposal.

Conclusion:

This study aims to provide evidence on the efficacy and safety of plasma transfusion in managing coagulopathy in non-bleeding thrombocytopenic dengue patients. Positive findings could lead to the incorporation of plasma transfusion into the standard care protocols, potentially improving patient outcomes in dengue-endemic regions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with dengue fever, thrombocytopenia (platelet count < 100,000/μL), and elevated aPTT (> 40 seconds) without active bleeding.

Exclusion Criteria:

* Patients with active bleeding, known coagulopathies unrelated to dengue, or contraindications to plasma transfusion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in aPTT values from baseline to 24 and 48 hours post-transfusion. | 24 to 48 hours
  Platelet count change from baseline (pre-intervention) to 48 hours post-transfusion. CBCs will be performed before FFP administration and 24 and 48 hours post-transfusion to measure platelets. The purpose is to determine if fresh frozen plasma (FFP) enhances platelet count in dengue-related thrombocytopenia patients compared to usual therapy without FFP.

SECONDARY OUTCOMES:
Incidence of bleeding complications within 7 days post-transfusion, changes in other coagulation parameters (PT, fibrinogen levels) from baseline to 24 and 48 hours post-transfusion, platelet count changes post-transfusion, length of hospital stay, and o | 30 days
  This outcome tracks hospitalized patients' minor and significant bleeding occurrences. Clinical severity will classify bleeding occurrences (e.g., petechiae, mucosal, gastrointestinal). Staff will collect data everyday through clinical assessments and record it in patient records. The experimental (FFP + standard care) and control (standard care alone) groups will be compared for bleeding problems.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraful Hoque, DBST, Principal Investigator — Sheikh Hasina National Institute of Burn & Plastic Surgery
Locations (1):
- SheikhHasinaNIBPS, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Yes
The researchers will have access to the de-identified individual participant data (IPD) that was collected during this trial upon a reasonable request. Individual participant data on baseline characteristics, primary and secondary outcome measures, and adverse event reports will comprise the shared data.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After 1st Novembar, 2024
Access Criteria: Access to de-identified individual participant data (IPD) will be granted to researchers who meet the following criteria:
  Scientifically Sound Proposal: Researchers must submit a valid scientific proposal outlining the objectives and methodology, subject to review by the study's steering committee.
  Ethics Approval: A valid ethics committee or IRB approval for secondary use of the data must be provided.
  Data Use Agreement (DUA): Researchers must sign a DUA ensuring data use is limited to approved purposes, maintains participant privacy, and follows data security measures.
  Non-commercial Use: Data access is limited to academic and public health research, not for commercial purposes.
  Publication: Researchers agree to publish their findings in peer-reviewed journals or other public formats.
  Security: Data must be handled in compliance with relevant privacy regulations.

REFERENCES:
- [Result] Lye DC, Lee VJ, Sun Y, Leo YS. Lack of efficacy of prophylactic platelet transfusion for severe thrombocytopenia in adults with acute uncomplicated dengue infection. Clin Infect Dis. 2009 May 1;48(9):1262-5. doi: 10.1086/597773. PMID 19292665
- [Result] Wills BA, Oragui EE, Dung NM, Loan HT, Chau NV, Farrar JJ, Levin M. Size and charge characteristics of the protein leak in dengue shock syndrome. J Infect Dis. 2004 Aug 15;190(4):810-8. doi: 10.1086/422754. Epub 2004 Jul 19. PMID 15272410
- [Result] Malavige GN, Velathanthiri VG, Wijewickrama ES, Fernando S, Jayaratne SD, Aaskov J, Seneviratne SL. Patterns of disease among adults hospitalized with dengue infections. QJM. 2006 May;99(5):299-305. doi: 10.1093/qjmed/hcl039. Epub 2006 Apr 7. PMID 16603571
- [Result] Martina BE, Koraka P, Osterhaus AD. Dengue virus pathogenesis: an integrated view. Clin Microbiol Rev. 2009 Oct;22(4):564-81. doi: 10.1128/CMR.00035-09. PMID 19822889
- [Result] Mackenzie JS, Gubler DJ, Petersen LR. Emerging flaviviruses: the spread and resurgence of Japanese encephalitis, West Nile and dengue viruses. Nat Med. 2004 Dec;10(12 Suppl):S98-109. doi: 10.1038/nm1144. PMID 15577938
- [Result] Bhatt S, Gething PW, Brady OJ, Messina JP, Farlow AW, Moyes CL, Drake JM, Brownstein JS, Hoen AG, Sankoh O, Myers MF, George DB, Jaenisch T, Wint GR, Simmons CP, Scott TW, Farrar JJ, Hay SI. The global distribution and burden of dengue. Nature. 2013 Apr 25;496(7446):504-7. doi: 10.1038/nature12060. Epub 2013 Apr 7. PMID 23563266
- [Result] Guzman MG, Harris E. Dengue. Lancet. 2015 Jan 31;385(9966):453-65. doi: 10.1016/S0140-6736(14)60572-9. Epub 2014 Sep 14. PMID 25230594
- [Result] undefined